CLINICAL TRIAL: NCT06552208
Title: Elaboration of a Prognostic Score Based on Patients With Malignant Biliary Obstruction
Brief Title: Biliary Obstruction of Neoplastic Origin Treated With Drainage. A Prognostic Study.
Acronym: PROBILI
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC18.0197 - PROBILI
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Malignant Biliary Obstruction
Keywords: Prognostic score; Biliary drainage; 30-day survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inclusion of patients with biliary drainage for inoperable malignant biliary obstruction and analysis of clinico-biological parameters

DETAILED DESCRIPTION:
All patients who had biliary drainage between April 1, 2014 and August 31, 2018 for inoperable malignant biliary obstruction will be included.

Clinical and biological baseline data will be recorded retrospectively. From the electronic medical records (M-Eva software), the following clinical data will be retrieved on the day of procedure: age, gender, body mass index (BMI), percentage of weight loss in the last three months, American Society of Anesthesiologists score (ASA) , Charlson score, Eastern Cooperative Oncology Group Performans Status (ECOG PS), comorbidities, cancer type, liver metastases, obstruction level, pre-procedural sepsis, type of procedure and type of stent.

Serum biological parameters will be recorded: hemoglobin, platelets, leukocytes, urea, creatinine, albumin, total bilirubin and prothrombin time, within 48 hours prior to the procedure.

The continuous variables of biological tests will be analyzed by ROC curves. The survival curves will be estimated using the Kaplan-Meier method and compared using the log-rank test. A prognostic index will be established from the variables independently associated with poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Malignant Biliary obstruction : cholestasis (elevated bilirubin > 40 µmol/L or alkaline phosphatase > 1.5 time than the normal value) and dilation of biliary tract

Exclusion Criteria:

* Benign obstruction
* Post stent surgery
* First stent placed outside Brest University Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohort will be selected from the general population of Brest, Finistère.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Short-term survival after biliary drainage | 4 years and fifth months
  30-day survival after biliary drainage

SECONDARY OUTCOMES:
Prognostic score | 4 years and fifth months
  To establish a prognostic score

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending three years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.